CLINICAL TRIAL: NCT05297825
Title: Twins Nutrition Study (TwiNS): Vegan vs. Omnivore
Acronym: TwiNS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Christopher Gardner, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 63995
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2023-12

CONDITIONS: Lipid Metabolism; Glucose Intolerance; Weight Change, Body; Microbiome; Inflammation; Immune Function
Keywords: Lipids; Glucose; Body weight; Microbiome; Inflammation; Immune function
MeSH Terms: conditions — Glucose Intolerance; Body Weight Changes; Inflammation; Body Weight | interventions — Diet, Vegan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vegan (Experimental): Participants will be asked to consume a healthy vegan diet.
  Interventions: Behavioral: Vegan diet
- Omnivore (Experimental): Participants will be asked to consume a healthy omnivore diet.
  Interventions: Behavioral: Omnivore diet

INTERVENTIONS:
Behavioral: Vegan diet — Healthy vegan diet.
  Arms: Vegan
Behavioral: Omnivore diet — Healthy omnivore diet.
  Arms: Omnivore

SUMMARY:
This study is designed to investigate the health impact of a vegan diet compared to a usual, omnivorous diet. The investigators plan to study these diets in twins, where one twin follows a vegan diet and the other twin follows an omnivorous diet, thus the investigators control for genetic differences that might impact the effect of the diet.

DETAILED DESCRIPTION:
During this study, the investigators will evaluate the nutrient intake in both the vegan and the omnivorous diet. The investigators will also measure physiologic markers of health such as lipid levels, HbA1C, heart rate, and weight, and they will also look at the effect of the diets on the microbiota. In addition to measuring the effect of the diet, the investigators will monitor adherence to the diet, and survey participants on the ease/difficulty in following a vegan diet as well as their energy levels and sense of wellbeing. Thus, this study will help us better understand the health impact and feasibility of following a vegan diet. These results will be of much interest to the general public and the health care professionals.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* 1/2 of a pair of twins that will both be participating
* Willing to consume a plant-based diet (vegetables, fruit, whole grains, legumes, etc.)
* Willing to consume meat/eggs (beef, pork/sausage, chicken, eggs) >= 1 time a day
* Willing to consume dairy (milk, yogurt, cheese) >= 1 time a day

Exclusion Criteria:

* Weight < 110 lb
* BMI >= 40
* LDL-C > 190 mg/dL
* Systolic Blood Pressure > 160 mmHg OR Diastolic blood pressure > 90 mmHg
* Pregnant, lactating or planning to become pregnant during the course of the study.
* Use of any of the following drugs/supplements within the last 2 months:

  * systemic antibiotics, antifungals, antivirals or antiparasitics (intravenous, intramuscular, or oral);
  * corticosteroids (intravenous, intramuscular, oral, nasal or inhaled);
  * cytokines;
  * methotrexate or immunosuppressive cytotoxic agents.
* Chronic, clinically significant, or unstable (unresolved, requiring on-going changes to medical management or medication) pulmonary, cardiovascular, gastrointestinal, hepatic or renal functional abnormality, as determined by medical history, Type 1 diabetes, dialysis
* History of active cancer in the past 3 years except for squamous or basal cell carcinomas of the skin that have been medically managed by local excision
* Unstable dietary history as defined by major changes in diet during the previous month, where the subject has eliminated or significantly increased a major food group in the diet.
* Recent history of chronic excessive alcohol consumption defined as more than five 1.5-ounce servings of 80 proof distilled spirits, five 12-ounce servings of beer or five 5-ounce servings of wine per day; or > 14 drinks/week.
* Any confirmed or suspected condition/state of immunosuppression or immunodeficiency (primary or acquired) including HIV infection, multiple sclerosis and Graves' disease.
* Surgery of the GI tract, with the exception of cholecystectomy and appendectomy, in the past five years. Any major bowel resection at any time.
* Regular/frequent use of smoking or chewing tobacco, e-cigarettes, cigars or other nicotine-containing products
* Regular use of prescription opiate pain medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Difference in LDL cholesterol | Baseline and 8 weeks
  Difference in the 8-week change-from-baseline in LDL cholesterol between the vegan vs. omnivore diet groups

SECONDARY OUTCOMES:
Difference in triglycerides | Baseline and 8 weeks
  Difference in the 8-week change-from-baseline in triglycerides between the vegan vs. omnivore diet groups
Change in inflammatory markers | Baseline and 8 weeks
  Difference in the 8-week change-from-baseline in inflammatory markers detected in blood samples between the vegan vs. omnivore diet groups.
Change in alpha diversity | Baseline and 8 weeks
  Change from baseline in alpha diversity at 8 weeks in the vegan and omnivore diet groups. We will be using the number of observed sequence variants ("species") determined by standard 16S rRNA amplicon sequencing (V3-V5 region followed by DADA2 to define error-corrected sequence variants) as our primary metric of alpha diversity. We will also determine whether there is a change in observed sequence variants between the two groups. Higher alpha diversity is better. The units are the number of sequence variants.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D Garnder, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Landry MJ, Ward CP, Cunanan KM, Durand LR, Perelman D, Robinson JL, Hennings T, Koh L, Dant C, Zeitlin A, Ebel ER, Sonnenburg ED, Sonnenburg JL, Gardner CD. Cardiometabolic Effects of Omnivorous vs Vegan Diets in Identical Twins: A Randomized Clinical Trial. JAMA Netw Open. 2023 Nov 1;6(11):e2344457. doi: 10.1001/jamanetworkopen.2023.44457. PMID 38032644
- [Derived] Zeitlin AB, Ward CP, Minerva Cooper AO, Landry MJ, Krenek AM, Durand LR, Cunanan KM, Robinson JL, Dant CC, Gardner CD. Diet Quality and Comparison of Plant-Based Versus Omnivore Diets in Identical Twins: A Secondary Analysis of the Twins Nutrition Study (TwiNS). Curr Dev Nutr. 2025 Sep 4;9(10):107549. doi: 10.1016/j.cdnut.2025.107549. eCollection 2025 Oct. PMID 41081008
- [Derived] Dwaraka VB, Aronica L, Carreras-Gallo N, Robinson JL, Hennings T, Carter MM, Corley MJ, Lin A, Turner L, Smith R, Mendez TL, Went H, Ebel ER, Sonnenburg ED, Sonnenburg JL, Gardner CD. Unveiling the epigenetic impact of vegan vs. omnivorous diets on aging: insights from the Twins Nutrition Study (TwiNS). BMC Med. 2024 Jul 29;22(1):301. doi: 10.1186/s12916-024-03513-w. PMID 39069614
- See also: Study description — https://med.stanford.edu/nutrition/research/completed-studies/twins.html